CLINICAL TRIAL: NCT06005558
Title: Comparative Study Between High and Low Dose Methylene Blue Infusion in Septic Cancer Patients. A Randomized Blinded Controlled Study
Brief Title: Low Dose Versus High Dose Methylene Blue in Septic Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, Associate Professor of Anesthesia, ICU and Pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Methylene blue
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Saline Solution; Methylene Blue; Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal saline (Active Comparator): 30 patients will receive placebo of 100ml 0.9% Nacl over 20 minutes followed by continuous infusion of Nacl for 72 hours.
  Interventions: Drug: Methylene Blue low dose; Drug: Methylene Blue high dose
- methylene blue low dose (Active Comparator): 30 patients will receive a bolus of MB 1mg/kg in 100ml 0.9% Nacl over 20 minutes followed by continuous infusion of 0.25mg/kg/hour for 72 hours.
  Interventions: Drug: Normal saline; Drug: Methylene Blue high dose
- methylene blue high dose (Active Comparator): 30 patients will receive a bolus of MB 4mg/kg in 100ml 0.9% Nacl over 20 minutes followed by continuous infusion of 0.25mg/kg/hour for 72 hours.
  Interventions: Drug: Normal saline; Drug: Methylene Blue low dose

INTERVENTIONS:
Drug: Normal saline — 100 ml 0.9% Nacl over 20 minutes, followed by continuous infusion of normal saline for 72 hours.
  Other Names: Control
  Arms: methylene blue high dose; methylene blue low dose
Drug: Methylene Blue low dose — A bolus of MB 1mg/kg in 100ml 0.9% Nacl over 20 minutes followed by continuous infusion of 0.25mg/kg/hour for 72 hours.
  Other Names: Low dose
  Arms: Normal saline; methylene blue high dose
Drug: Methylene Blue high dose — A bolus of MB 4mg/kg in 100ml 0.9% Nacl over 20 minutes followed by continuous infusion of 0.25mg/kg/hour for 72 hours.
  Other Names: High dose
  Arms: Normal saline; methylene blue low dose

SUMMARY:
The main aim of this study is to examine the various effects of continuous methylene blue infusion in septic cancer patients and to compare it with the traditional infusion of noradrenaline in such patients .

DETAILED DESCRIPTION:
Exaggerated host response to infection, may result in sepsis, which is life-threatening organ dysfunction . Though considered the number one cause of in-hospital deaths , it can be treatable with early prompt interventions.

The 2021 SSC Guidelines use the Third International Consensus definitions, also known as Sepsis-3. Where sepsis is defined as "life-threatening organ dysfunction caused by a dysregulated host response to infection." Organ dysfunction is evidenced by an increased score of 2 or more in the Quick Sequential [Sepsis-related] Organ Failure Assessment (QSOFA), and septic shock is considered as "a subset of sepsis in which particularly profound circulatory, cellular, and metabolic abnormalities are associated with a greater risk of mortality than with sepsis alone." To diagnose septic shock, an euvolemic patient must require vasopressor support to achieve a mean arterial pressure of at least 65 mm Hg and have a lactate level above 2 mmol/L.

The triad of intravenous fluid, vasopressors and antibiotics in the first hour is the mainstay of septic shock management. Aim of management is to maintain patient hemodynamically stable until antibiotics kick in and fight infection. In case of non-responders, low dose corticosteroids are prescribed. Other drugs need to be studied to also help in cases of non-responders and to improve outcome in general. Methylene blue (MB) is a nitric oxide inhibitor that can counteract the vasodilatation in early septic shock.

Nitric oxide (NO) activates soluble guanylyl cyclase (sGC) which activates cyclic guanosine monophosphate (cGMP)-dependent protein kinases (PKGs) that cause vasodilatation. Methylene blue selectively blocks sGC and inhibits iNOS. Therefore, it selectively acts on the microcirculation.

Onset of action of intravenous MB is 30-60 min. Peak concentration at 30 min. It is excreted through bile and fecal routes plus through the kidneys. Due to the short Plasma half-life of 5-6 hours, some studies used continuous infusion of 0.25-2 mg/kg/h, for up to 3 days following the initial bolus dose

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years and ≤ 65 with septic shock as defined by Sepsis-3 criteria (confirmed infection, requiring vasopressor to maintain a mean arterial blood pressure (MAP) ≥ 65 mmHg, and serum lactate > 2 mmol/L after adequate fluid resuscitation), and requiring mechanical ventilation.

Exclusion Criteria:

* myocardial infarction or cerebrovascular accident within the last 3 months.
* severe lung , liver or kidney disease (creatinine >3.5 mg/dL).
* pregnancy.
* glucose 6-phosphate-dehydrogenase deficiency.
* known allergy to MB or food dyes and the use of nitrates within the last 3 days.
* more than 24 hrs since initiation of norepinephrine.
* other causes of shock than sepsis .
* recent intake (4-weeks) of selective serotonin re-uptake inhibitors or MAOi.
* refusal of the patient guardian to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Discontinuation of vasopressor | 7 days
  Time for noradrenaline discontinuation

SECONDARY OUTCOMES:
Mortality | 28 days
  Number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Shaker, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
After study completion and study publication we can share IPD upon request.

REFERENCES:
- [Result] Chalise SN, Sahib TA, Boyer GA, Pathak V. Methylene Blue in Refractory Shock. Cureus. 2022 Nov 6;14(11):e31158. doi: 10.7759/cureus.31158. eCollection 2022 Nov. PMID 36505110
- [Derived] Shaker EH, Soliman AM, Bedewy AAE, Elrawas MM. Comparative study between high and low dose methylene blue infusion in septic cancer patients: a randomized, blinded, controlled study. BMC Anesthesiol. 2025 Jan 8;25(1):15. doi: 10.1186/s12871-024-02792-3. PMID 39780053